CLINICAL TRIAL: NCT02581605
Title: Patient Matched Osteotomy to Correct Angular Deformities in Knee Arthrosis
Brief Title: Correction of Angular Deformities in Knee Arthrosis
Status: Active, not recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 13/LO/1639
Record Dates: First submitted 2015-09-21; First posted 2015-10-21 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Arthritis of Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Osteotomy Arm: Patients due to undergo an osteotomy around the knee. To improve the accuracy of this operation we propose the use of a custom-made 'cutting block' tailored for each individual patient.
  Interventions: Device: Custom-made 'cutting block'
- Partial Knee Replacement Arm: Patients due to undergo a partial knee replacement. To improve the accuracy of this operation we propose the use of a custom-made 'cutting block' tailored for each individual patient.
  Interventions: Device: Custom-made 'cutting block'

INTERVENTIONS:
Device: Custom-made 'cutting block' — To improve the accuracy of this operation we propose the use of a custom-made 'cutting block' tailored for each individual patient.

SUMMARY:
For participants whose leg bones don't line up properly, extra stress is placed on either the inner or outer side of the knee joint due to uneven transfer of body-weight. Gradually, this extra pressure wears away the smooth cartilage, resulting in osteoarthritis on that side of the knee joint. This problem is particularly common in young athletes and places them at risk of early osteoarthritis.

An operation exists whereby one of the bones either side of the knee is cut ( an osteotomy) and hinged open to straighten the leg. This alteration redistributes body-weight more equally across the knee joint and is known to be effective in delaying and possibly preventing, the progression of knee osteoarthritis- especially in younger and physically more active patients in whom a knee replacement is undesirable.

Currently it is possible to ( accurately) calculate the precise position of the bone cut and number of degrees correction required to straighten a leg using digital x-rays and three-dimensional CT scans. However there is no method of implementing this pre-operative plan during surgery so that the majority of surgeons rely on relatively crude and ipso facto unreliable intra-operative measurements as a guide.

To improve the accuracy of this operation, the investigator propose the use of a custom-made 'cutting block', tailored for each individual patient and its shape will match the contour of the patient's bone to ensure it can only be placed in one position. Pre-cut slots and holes will then guide the saw cut and the number of degrees the bone in hinged open, as per the pre-operative plan; it functions as an intra-operative template for the surgeon.

This study will primarily examine whether there is a close match between the planned and actual correction of leg deformities when using a patient-matched cutting-block.

DETAILED DESCRIPTION:
Malalignment of the leg is known to play a significant role in the development of knee arthrosis. Osteotomy can be used to correct angular deformities around the knee. A number of studies have found that the success of this procedure in delaying the progression of knee arthrosis is highly dependent on an accurate of deformity correction.

It is possible to produce a precise pre-operative surgical plan of the osteotomy required for a favourable outcome. However, the majority of surgeons still rely upon relatively crude and ipso facto unreliable intra-operative measurements to guide the actual operation. This is reflected in studies comparing the pre-operative plan with final outcome.

So to facilitate accurate translation of pre-operative osteotomy planning to intra-operative execution, the investigator proposes to transfer two technologies that are already commercially available in arthroplasty into the filed of corrective osteotomy i.e. 3D planning and custom-made patient-matched cutting blocks. This will permit translation of the surgeon's pre-order to ensure precise intra-operative positioning. Once secured slots and holes in the cutting block will ensure that the bony cut and angular correction is performed, and secured with a plate and screws, in the precise location determined by the pre-operative plan.

A prospective multi centre study is proposed, primarily to confirm the efficacy of use, and accuracy of deformity correction around the knee using patient-matched cutting blocks. Accuracy will be assessed by comparing post-operative alignment (measured on plan radiographs and CT scan) with the pre-operative surgical plan. Patient questionnaires to assess outcome will also be collected, and optional gait analysis performed.

ELIGIBILITY:
Osteotomy Arm

Inclusion Criteria:

* All patients considered suitable candidates for an osteotomy around the knee.
* All patients consenting to an osteotomy around the knee.
* All patients considered medically fit for surgery.
* All patients must be between 18 to 70 years of age.

Exclusion Criteria:

* Patients not suitable for an osteotomy around the knee.
* Patients with collateral ligament(s) insufficiency.
* Patients who decline surgery.
* Patients lacking capacity to consent.
* Patients who do not understand English (written and verbal).

Partial Knee Replacement Arm:

Inclusion Criteria

* All patients considered suitable candidates for a partial knee replacement
* All patients consenting to a partial knee replacement
* All patients considered medically fit for surgery Exclusion Criteria
* Patients not suitable for a partial knee replacement.
* Patients who decline surgery.
* Patients lacking capacity to consent.
* Patients under the age of eighteen.
* Patients who do not understand English (written and verbal).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Osteotomy Arm:
  Target population: 42
  Partial Knee Replacement Arm:
  Target population: 42
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2014-11; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Final radiographic alignment is with two degrees of pre-operative plan in both coronal and sagittal | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Professor Justin Cobb, Principal Investigator — Imperial College London
Locations (1):
- Charing Cross Hospital, London, United Kingdom